CLINICAL TRIAL: NCT02633618
Title: The Clinical Study of Analgecine for the Treatment of Neuropathic Pain
Brief Title: Analgecine for the Treatment of Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VanWorld Pharmaceutical (Rugao) Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004L04536
Record Dates: First submitted 2015-11-30; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — neurotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Analgecine (Experimental): 3ml, 2 times per day, continuous infusion for two weeks.
  Interventions: Biological: Analgecine
- Neurotropin (Active Comparator): 3ml, 2 times per day, continuous infusion for two weeks.
  Interventions: Biological: Neurotropin

INTERVENTIONS:
Biological: Analgecine — Extraction from rabbit skin extract through vaccinia virus inoculation inflammation as an antigen immune reaction.
  Arms: Analgecine
Biological: Neurotropin — a natural bio-product obtained from rabbit skin extract through vaccinia virus inoculation inflammation as an antigen immune reaction.
  Arms: Neurotropin

SUMMARY:
A randomized, open-label , positive drug controlled (Neurotropin,Japan organs Pharmaceutical Co., Ltd. ), multi-center study to evaluate Analgecine's efficacy and safety for the treatment of neuropathic pain.

DETAILED DESCRIPTION:
The study was designed to evaluate the efficacy and safety of Analgecine for the treatment of neuropathic pain for 2 weeks. It was a randomized, open-label , positive drug controlled, multi-center study phase III clinical trial. Patients were recruited with age between 18 and 80 and visual analysis scale (VAS) between 3 and 8. After randomization, subjects were divided into 2 groups: 1) Treatment with Analgecine as experiment group; 2) Treatment with Neurotropin as positive control group. There are 3 measurement time points on day 0, 7, 14 after treatment to score patients pain with VAS. The changes of the VAS score at day 14 were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the established medical records;
2. Patients with age of 18 years to 80 years old.
3. Patients with neuropathic pain
4. Patients at child-bearing age with negative pregnancy tests and contraceptive measures ( oral or injectable contraceptives) taken throughout the course of the experiment
5. Patients with signed informed consent.

Exclusion Criteria:

1. Patients younger than 18 years old or older 80 years old
2. Patients of dementia who can not determine efficacy
3. Patients who was pregnant, nursing or who may become pregnant in the study course and did not take effective contraceptive measures.
4. Patients with the history of allergic reactions
5. Patients suffering from tuberculosis, cancer and other organic disease
6. Patients who are alcoholics and drug addicts
7. Others who were determined by physician not to be a candidate for this clinical observation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2005-08; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change of visual analog scale on pain | 2 weeks
  Pain was scored by VAS 10 points (visual analog scale). The degree of pain gradually increases from 0 to 10. The subtraction mark rate of VAS value before and after treatment and the grade decrease of associated symptoms will be regarded as the main curative effects indexes.

CONTACTS AND LOCATIONS:
Overall Officials: Lu-Ning Wang, Study Director — Chinese PLA General Hospital